CLINICAL TRIAL: NCT01226108
Title: The Akloma Tinnitus Patch in Patients With Manifested Tinnitus (the Aktin Study)
Brief Title: The Akloma Tinnitus Patch in Patients With Manifested Tinnitus
Acronym: Aktin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akloma Bioscience AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Aktin study
Record Dates: First submitted 2010-10-20; First posted 2010-10-21 (Estimated); Last update posted 2011-09-26 (Estimated); Status verified 2011-09

CONDITIONS: Tinnitus
MeSH Terms: conditions — Tinnitus | interventions — Transdermal Patch

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- antinitus patch (Active Comparator): One patch per day, Duration: three weeks, Administration: behind the ear
  Interventions: Device: Patch

INTERVENTIONS:
Device: Patch — One patch per day, Duration: three weeks, Administration: behind the ear
  --------------------------------------------------------------------------------

SUMMARY:
OBJECTIVES:

Primary Objective The primary objective will be a decrease of inconvenience with at least 10% for at least 50% of the subjects.

Secondary Objectives

The secondary objective will be to:

To evaluate if the patch can improve the tinnitus patient's quality of life and sleep quality.

METHODOLOGY

Study Design:

An open safety and performance clinical investigation of the antinitus patch in patients with manifested tinnitus.

Treatment Duration:

1 patch per day for 3 weeks

Primary Endpoint:

Tinnitus severity questionnaire (TSQ)

Performance Parameters:

Tinnitus severity questionnaire (TSQ) and numerical rating scale (NRS) measuring tinnitus annoyance.

Quality of life and sleep quality

Safety Parameters: Adverse Reactions

ELIGIBILITY:
Inclusion Criteria:

* Adults of both sexes > 18 years of age
* Signed informed consent
* Patients who have suffered from tinnitus for ≥ 4 weeks before study entry
* Manifested tinnitus grade II or above on the Klockhoff-Lindblom tinnitus severity grading scale.
* Tinnitus score of 5 or above (numerical rating scale for tinnitus annoyance)
* Pure tone averages better than 40 dB in the worse hearing ear.

Exclusion Criteria:

* Pregnant or lactating women
* Malignancy or other serious medical conditions
* Skin disease
* Simultaneous or previous (within 30 days prior to study entry) participation in a clinical study using experimental drugs or devices.
* Severe psychiatric disorder
* Serious suicidal risk
* Patients who have started treatment or made changes in treatment with drugs known to influence tinnitus within 6 weeks before study start.
* Patients with untreated high blood pressure ≥140/90 mmHg
* Other tinnitus treatment within 6 weeks before study entry.
* Previous use of the Antinitus patch
* Known allergy or sensitivity to any of the compounds in the Antinitus or the placebo patches.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2010-10; Primary Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 7 weeks
Tinnitus severity questionnaire score as a measure of efficacy | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Peter Åhnblad, Principal Investigator — Sickla ÖNH-center / Supramed AB
Locations (1):
- Sickla ÖNH-center, Atlashuset Planiavägen 5, Nacka, Sweden